CLINICAL TRIAL: NCT06024291
Title: Reducing Circulating Sphingolipid Levels to Optimise Cardiometabolic Health - The SphingoFIT Randomised Controlled Exercise Trial
Brief Title: Reducing Circulating Sphingolipid Levels to Optimise Cardiometabolic Health - The SphingoFIT Trial
Acronym: SphingoFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: University of Lausanne (Other); Technical University of Munich (Other)
Responsible Party: Principal Investigator, Justin Carrard, Postdoctoral researcher, Principal investigator, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EKNZ 2023-01345
Record Dates: First submitted 2023-08-28; First posted 2023-09-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Overweight and Obesity; Dyslipidemias; Blood Pressure; Cardiovascular Diseases; Metabolic Disease
MeSH Terms: conditions — Overweight; Obesity; Dyslipidemias; Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: As the randomisation will take place after the baseline examination, participants, exercise scientists, and physicians supervising the intervention will be blinded for group allocation at baseline but not post-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIIT group (Experimental): The exercise intervention will consist of a supervised HIIT (two walking- and one indoor cycling-based session weekly), starting with a habituation week at an intensity of 75% of the maximal heart rate (HRmax). In the following seven weeks, the participants will perform a HIIT based on the following protocol and for a total duration of 45 min per session: warm-up for 10 min at 60%-70% HRmax followed by a high-intensity interval consisting of 4×4 min at 80%-95% HRmax with 3 min of active recovery at 60%-70% HRmax and a 10 min cool-down at 60%-70% HRmax. Heart rate will be monitored during training by Garmin HRM-Dual heart rate sensors combined with Garmin Forerunner 45S watches. Exercise scientists motivate the participants during the intervals and will control each participant's heart rate during and after every training session.
  Interventions: Other: 8-week HIIT programme
- Physical activity recommendation group (Active Comparator): Asking physically inactive participants to maintain their inactive habits may not reflect realistic conditions and is no longer considered the best option in a randomised controlled exercise intervention. Indeed, most participants will be aware of the positive effects of PA - or will become aware of them during an exercise intervention study. Further, denying an exercise intervention to participants who would have benefited from it (for instance, participants at risk of cardiometabolic diseases) might be ethically questionable. In accordance with current practices, control group participants will be informed about the World Health Organization physical activity guidelines at the beginning of the study.
  Interventions: Other: Physical activity recommendation

INTERVENTIONS:
Other: 8-week HIIT programme — See arm description
  Arms: HIIT group
Other: Physical activity recommendation — See arm description
  Arms: Physical activity recommendation group

SUMMARY:
The purpose of this study is to assess the effects of an 8-week supervised high-intensity interval training (HIIT) program (vs. physical activity recommendations according to current guidelines) on a comprehensive panel of circulating sphingolipids in middle-aged females and males at elevated cardiometabolic risk.

DETAILED DESCRIPTION:
Cardiometabolic diseases (CMD) account for about half of all deaths from non-communicable diseases and are responsible for about one-third of all deaths worldwide. To combat the growing burden of CMD on health systems, a shift towards more effective prevention and early detection of these diseases is urgently needed.

Blood lipids have been used since the middle of the last century to determine the risk of developing CMD. Although classically used biomarkers such as cholesterol and triglycerides provide acceptable risk assessment, there is increasing evidence that sphingolipids, particularly ceramides, may allow improved risk assessment. Mechanistically, there is growing data that sphingolipid accumulations lead to atherosclerosis and insulin resistance.

To measure circulating sphingolipids in clinical practice, it is essential to provide patients with evidence-based interventions that reduce sphingolipid levels and quantify the reduction expected from such an intervention. Preliminary data suggest that regular physical activity (PA), an effective, low-cost, and patient-empowering means of health optimisation, may reduce sphingolipid levels.

The current research project aims to explore whether and to what extent a fitness-enhancing high-intensity interval training (HIIT) programme can lower circulating sphingolipid levels in middle-aged individuals at elevated cardiometabolic risk (50% females). An 'omic-scale sphingolipid profiling will be applied to capture the circulating sphingolipidome comprehensively.

Participants will be randomly allocated to either the intervention or the control group. The exercise intervention will consist of an 8-week supervised HIIT (two walking- and one indoor cycling-based session weekly). The control group will get PA recommendations based on current guidelines.

Maximal cardiopulmonary exercise testing (CPET) will be conducted on a cycle ergometer to determine the VO2peak, peak heart rate and peak power output. After the 8-week training programme, a second CPET will be performed to verify if the exercise intervention effectively improved CRF. Body composition will be analysed before and after the 8-week intervention by dual-energy x-ray absorptiometry and by bioelectrical impedance analysis.

Trained medical staff will draw blood samples by venepuncture of the cubital fossa following an overnight fast pre- and post-intervention. Planned blood analyses for basic characterisation of risk factor profiles include total cholesterol, low-density lipoprotein cholesterol (LDL) and high-density lipoprotein cholesterol (LDL), triglycerides, and HbA1c. Glucose and insulin will also be measured to estimate insulin resistance using the HOMA-IR. A high-coverage method using reversed-phase liquid chromatography coupled to tandem mass spectrometry (RPLC-MS/MS) will be applied to quantify an extensive panel of circulating sphingolipids (n=61).

Retinal vessel diameters, a novel surrogate of microvascular health that responds positively to exercise interventions, will be assessed pre- and post-intervention, and the brachial artery FMD, which reflects endothelial function as an early marker of atherosclerotic arterial damage.

Each participant will receive individualised, pre-packaged meals for the two days preceding blood sampling to minimise potential confounding. All participants will be fed to energy balance. To monitor diet adherence, participants will be instructed to return all non-consumed foods from the pre-packaged meals to the lab and take photos of additionally consumed foods for later analysis.

ELIGIBILITY:
Inclusion Criteria:

* female or male sex,
* aged between 40 and 60 years,
* body mass index between 25.0 and 34.9 kg/m2,
* sedentary lifestyle, defined as not meeting the WHO guidelines on PA, i.e., at least 150 minutes of moderate-intensity aerobic PA per week as well as muscle-strengthening activities on two or more days per week,
* medical clearance for HIIT by a study physician (including vital sign evaluation, clinical examination, resting and exercise ECG),
* informed consent as documented by signature.

Exclusion Criteria:

* known pregnancy or breastfeeding,
* any current exercise-limiting musculoskeletal conditions of the lower limbs,
* any known current or chronic conditions limiting exhaustive exercise,
* known diabetes mellitus of any type,
* dyslipidaemia, if pharmaceutically treated,
* arterial hypertension ≥160/100 mmHg, pharmaceutically treated or not,
* any other known cardiovascular disease,
* known NASH,
* known macular degeneration, glaucoma, or high intraocular pressure (≥20 mm Hg),
* particular diet (vegetarian, vegan, lactose-free, gluten-free, or FODMAP-low diet (ferment-able oligosaccharides, disaccharides, monosaccharides, and polyols),
* intake of glucagon-like peptide-1 analogues, orlistat or any weight-loss drug,
* inability to follow the procedures of the study, e.g., due to linguistic or cognitive problems,
* concomitant involvement in another interventional trial or participation in another interventional trial in the last four weeks.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Concentration of circulating Cer16:0, Cer18:0, Cer24:0 and Cer24:1 | At baseline and after the 8-week intervention
  Quantifying the changes in plasma level of the four sphingolipid species included in the ceramide-based scores (Cer16:0, Cer18:0, Cer24:0 and Cer24:1) following the 8-week HIIT programme (vs. physical activity recommendation).

SECONDARY OUTCOMES:
Concentration of the other circulating sphingolipid species to be targeted | At baseline and after the 8-week intervention
  Quantifying the changes in plasma level of the other sphingolipids to be targeted following the 8-week HIIT programme (vs. physical activity recommendation).
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | At baseline and after the 8-week intervention
  Quantifying the changes in HOMA-IR following the 8-week HIIT programme (vs. physical activity recommendation).
Peak oxygen uptake (VO2peak) | At baseline and after the 8-week intervention
  Quantifying the changes in VO2peak following the 8-week HIIT programme (vs. physical activity recommendation).
Retinal microvascular diameters | At baseline and after the 8-week intervention
  Quantifying the changes in retinal microvascular diameters following the 8-week HIIT programme (vs. physical activity recommendation).
Brachial flow-mediated dilatation (FMD) | At baseline and after the 8-week intervention
  Quantifying the changes in FMD following the 8-week HIIT programme (vs. physical activity recommendation).

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, Prof, MD, MA, Study Chair — Department of Sport, Exercise and Health, University of Basel, Basel, Switzerland
Locations (1):
- Department of Sport, Exercise and Health, University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi RH, Tatum SM, Symons JD, Summers SA, Holland WL. Ceramides and other sphingolipids as drivers of cardiovascular disease. Nat Rev Cardiol. 2021 Oct;18(10):701-711. doi: 10.1038/s41569-021-00536-1. Epub 2021 Mar 26. PMID 33772258
- [Background] Laaksonen R, Ekroos K, Sysi-Aho M, Hilvo M, Vihervaara T, Kauhanen D, Suoniemi M, Hurme R, Marz W, Scharnagl H, Stojakovic T, Vlachopoulou E, Lokki ML, Nieminen MS, Klingenberg R, Matter CM, Hornemann T, Juni P, Rodondi N, Raber L, Windecker S, Gencer B, Pedersen ER, Tell GS, Nygard O, Mach F, Sinisalo J, Luscher TF. Plasma ceramides predict cardiovascular death in patients with stable coronary artery disease and acute coronary syndromes beyond LDL-cholesterol. Eur Heart J. 2016 Jul 1;37(25):1967-76. doi: 10.1093/eurheartj/ehw148. Epub 2016 Apr 28. PMID 27125947
- [Background] Tippetts TS, Holland WL, Summers SA. Cholesterol - the devil you know; ceramide - the devil you don't. Trends Pharmacol Sci. 2021 Dec;42(12):1082-1095. doi: 10.1016/j.tips.2021.10.001. Epub 2021 Nov 5. PMID 34750017
- [Background] Carrard J, Angst T, Weber N, Bienvenue J, Infanger D, Streese L, Hinrichs T, Croci I, Schmied C, Gallart-Ayala H, Hochsmann C, Koehler K, Hanssen H, Ivanisevic J, Schmidt-Trucksass A. Investigating the circulating sphingolipidome response to a single high-intensity interval training session within healthy females and males in their twenties (SphingoHIIT): Protocol for a randomised controlled trial. F1000Res. 2023 Aug 18;11:1565. doi: 10.12688/f1000research.128978.3. eCollection 2022. PMID 37533665
- [Derived] Carrard J, Hofer M, Prechtl L, Fleischlin E, Huber M, Gallart-Ayala H, Teav T, Infanger D, Hochsmann C, Koehler K, Hinrichs T, Hanssen H, Ivanisevic J, Schmidt-Trucksass A. Effect of an eight-week high-intensity interval training programme on circulating sphingolipid levels in middle-aged adults at elevated cardiometabolic risk (SphingoFIT)-Protocol for a randomised controlled exercise trial. PLoS One. 2024 May 8;19(5):e0302477. doi: 10.1371/journal.pone.0302477. eCollection 2024. PMID 38717997